CLINICAL TRIAL: NCT04291040
Title: Use of an Educational Multimedia Tool Versus Routine Care for the Uptake of Postpartum LARC in High-Risk Pregnancies (SUSTAIN): A Randomized Clinical Trial
Brief Title: Use of an Educational Multimedia Tool Versus Routine Care for the Uptake of Postpartum LARC in High-Risk Pregnancies
Acronym: SUSTAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Emma Jean Qureshey, Clinical MFM Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-20-0022
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy, High Risk; Contraception
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decision Aid (Experimental)
  Interventions: Behavioral: Decision Aid
- Routine Care (Active Comparator)
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Decision Aid — Following randomization, participants will independently view the multimedia based decision aid on a provided tablet. They will also receive provider counseling. For the remainder of the pregnancy, they will receive a text message with a link to the multimedia based presentation. This will occur every 4 weeks until 12 weeks postpartum.
  Arms: Decision Aid
Behavioral: Routine Care — The control arm will receive routine prenatal care including provider counselling on postpartum contraceptive options.
  Arms: Routine Care

SUMMARY:
The purpose of the study is to evaluate if the implementation of a multimedia based educational tool and regular reminders with shared decision-making will increase the rate of LARC uptake and retention in high risk pregnancy patients within 12 weeks of delivery and to study the rates of retention of LARC at 12 and 24 months and short-interval pregnancy rates.

DETAILED DESCRIPTION:
This study will include 380 women aged 18-50 enrolled between 28 weeks gestation and postpartum day #1 who have a pregnancy that is considered high-risk. After consent, participants will be randomized to either routine care or multimedia based intervention. The intervention will include an investigator created decision aid presented at the time of randomization and reminder texts until 12 weeks postpartum.

The primary objective is to evaluate the rate of LARC uptake and retention within 12 weeks of delivery. Secondary objectives include i) the retention of LARC at 12 and 24 months and ii) short-interval pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-50 years old
* High risk pregnancy due to either maternal medical conditions or obstetric/neonatal complications

Exclusion Criteria:

* Planned cesarean hysterectomy
* Unable to provide informed consent in either English or Spanish
* Unable to provide reliable cell phone access for the study duration
* Not willing to provide follow-up for two years

Ages: 13 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 380 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Rate of initial LARC utilization | 12 weeks postpartum (12 weeks)
  Number of subjects who elect to have LARC procedure between the 2 arms

SECONDARY OUTCOMES:
Number of patients who keep the LARC after placement | 12 months
Number of patients who keep the LARC after placement | 24 months
rates of short interval pregnancy | 24 months
  Number of patients who become pregnant after enrollment pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qureshey EJ, Ibarra CJ, Wagner SM, Chen HY, Ashimi S, Ross PJ, Blackwell SC, Sibai BM, Chauhan SP. Effect of a Multimedia Educational Tool on Contraception Use 1 Year Postpartum. Obstet Gynecol. 2023 Jun 1;141(6):1206-1208. doi: 10.1097/AOG.0000000000005198. Epub 2023 May 3. PMID 37141601
- [Derived] Qureshey EJ, Chauhan SP, Wagner SM, Batiste O, Chen HY, Ashimi S, Ross PJ, Blackwell SC, Sibai BM. Educational Multimedia Tool Compared With Routine Care for the Uptake of Postpartum Long-Acting Reversible Contraception in Individuals With High-Risk Pregnancies: A Randomized Controlled Trial. Obstet Gynecol. 2022 Apr 1;139(4):571-578. doi: 10.1097/AOG.0000000000004718. Epub 2022 Mar 10. PMID 35594122